CLINICAL TRIAL: NCT03848741
Title: Independent and Combined Effects of Resistance Exercise Training and β-hydroxy β-methylbutyrate Plus Vitamin D on Body Composition and Skeletal Muscle Health
Brief Title: Independent and Combined Effects of Resistance Exercise Training and β-hydroxy β-methylbutyrate Plus Vitamin D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Metabolic Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Adam Konopka, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 093635
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Aging; Skeletal Muscle
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1 of 4, 12-week interventions. In a double-blinded fashion, participants will be randomized to consume either placebo or HMB + VitD supplementation.
  Group 1 will serve as a non-exercise control with placebo; Group 2 will serve as a non-exercise control with β-hydroxy β-methylbutyrate + Vitamin D; Group 3 will complete resistance exercise training with placebo; Group 4 will complete resistance exercise training with β-hydroxy β-methylbutyrate + Vitamin D
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-exercise control with placebo (Placebo Comparator): Participants will be asked to maintain their normal physical activity and dietary habits during the 12-week intervention. Physical activity, diet, urine and blood samples will be collected every 4 weeks. Each participant will consume 3 placebo capsules (calcium lactate), twice a day with a meal or snack for a total of 6 capsules per day. Placebo capsules match the size, color, weight, and number of capsules per dose compared to the β-hydroxy β-methylbutyrate (HMB) Plus Vitamin D (VitD) capsules.
  Interventions: Behavioral: Non-Exercise Control; Dietary Supplement: Placebo
- Non-exercise control with HMB+VitD (Experimental): Participants will be asked to maintain their normal physical activity and dietary habits during the 12-week intervention. Physical activity, diet, urine and blood samples will be collected every 4 weeks. Each participant will consume 3 HMB+VitD capsules, twice a day with a meal or snack for a total of 6 capsules per day. Each capsule contains 500 mg calcium HMB and 333.33 IU Vitamin D for a total of 3.0 g HMB and 2000 IU Vitamin D per day.
  Interventions: Behavioral: Non-Exercise Control; Dietary Supplement: HMB+VitD
- Resistance exercise training with placebo (Active Comparator): Participants will complete 12-weeks (3 days per week) of a whole-body progressive resistance exercise training program. Physical activity, diet, urine and blood samples will be collected every 4 weeks. Each participant will consume 3 placebo capsules (calcium lactate), twice a day with a meal or snack for a total of 6 capsules per day. Participants will be asked to take capsules ~30-60 minutes before resistance exercise. Placebo capsules match the size, color, weight, and number of capsules per dose compared to the HMB + VitD capsules.
  Interventions: Behavioral: Resistance Exercise Training; Dietary Supplement: Placebo
- Resistance exercise training with HMB+VitD (Experimental): Participants will complete 12-weeks (3 days per week) of a whole-body progressive resistance exercise training program. Physical activity, diet, urine and blood samples will be collected every 4 weeks. Each participant will consume 3 HMB+VitD capsules, twice a day with a meal or snack for a total of 6 capsules per day. Participants will be asked to take capsules ~30-60 minutes before resistance exercise. Each capsule contains 500 mg calcium HMB and 333.33 IU Vitamin D for a total of 3.0 g HMB and 2000 IU Vitamin D per day.
  Interventions: Behavioral: Resistance Exercise Training; Dietary Supplement: HMB+VitD

INTERVENTIONS:
Behavioral: Non-Exercise Control — Participants will not perform structured exercise and will continue with their normal physical activity for 12-weeks.
  Arms: Non-exercise control with HMB+VitD; Non-exercise control with placebo
Behavioral: Resistance Exercise Training — Participants will complete a 12-week whole-body progressive resistance exercise training program.
  Arms: Resistance exercise training with HMB+VitD; Resistance exercise training with placebo
Dietary Supplement: Placebo — Participants will be given placebo capsules to consume for 12-weeks.
  Arms: Non-exercise control with placebo; Resistance exercise training with placebo
Dietary Supplement: HMB+VitD — Participants will be given HMB+VitD capsules to consume for 12-weeks
  Arms: Non-exercise control with HMB+VitD; Resistance exercise training with HMB+VitD

SUMMARY:
During middle-age, humans begin to lose muscle mass and strength. With increasing age the deterioration of muscle health is associated with a decline in quality of life and the loss of independence. β-hydroxy β-methylbutyrate (HMB) plus Vitamin D (VitD) have been proposed to increase skeletal muscle mass, contractile function and improve body composition but has yet to be evaluated in middle-aged women. The overall goal of this study is to determine the effects of HMB +VitD supplementation during 12 weeks of resistance exercise training or a non-exercise control on body composition, skeletal muscle size, and skeletal muscle function in middle-aged women.

DETAILED DESCRIPTION:
To determine if HMB+VitD supplementation is an effective strategy to help prevent the loss of skeletal muscle size, skeletal muscle function and body composition in middle-aged women, forty eight women (45-60 yrs old) will be recruited to complete a 12-week intervention (n=12 per group; 4 groups). Participants will be randomized to complete a non-exercise control period or a resistance exercise training program. In a double-blinded fashion, participants in the non-exercise or resistance exercise groups will be randomized to consume either placebo or HMB+VitD. Before and after each intervention the investigators will evaluate skeletal muscle size, skeletal muscle function, and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Women between 45 and 60 years old
* Women with a BMI < 35 kg/m2
* Sedentary (< 30 minutes of structured physical activity 3 times per week)
* Weight stable for 3 months prior (+/- 5kg)

Exclusion Criteria:

* Body mass index > 35 kg/m2
* Type 1 or Type 2 diabetes
* Uncontrolled hypertension
* Active cancer, cancer in remission, or having received treatment for any form of cancer in the previous 5 years
* Cardiovascular disease (e.g., peripheral artery disease and peripheral vascular disease)
* Uncontrolled thyroid function
* Chronic and/or regular consumption of medication known to influence skeletal muscle metabolism
* Use of Vitamin D (>2000 IU) or β-hydroxy β-methylbutyrate
* Tobacco use
* Any condition that limits exercise training (e.g., chronic obstructive pulmonary disease, neuromuscular disorder, moderate or severe cognitive impairment, Alzheimer's disease, vertigo, dizziness)
* High alcohol consumption defined as more than 8 drinks per week for women
* Unwilling to undergo any study-related procedures
* Pregnancy
* Abnormal liver or kidney enzymes determined in blood chemistry panel
* Bleeding/clotting disorders or blood thinning medications (e.g., warfarin, heparin)

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Function - Knee extensor isometric performance | Change from baseline to after the 12 week intervention
  Knee extensor isometric performance will be assessed by a dynamometer. Muscle strength will also be determined by 1 repetition maximum for leg extension, leg curl and leg press exercises.
Skeletal Muscle Function - Knee extensor isokinetic performance | Change from baseline to after the 12 week intervention
  Knee extensor isokinetic performance will be assessed by a dynamometer.
Skeletal Muscle Function - Fatigue | Change from baseline to after the 12 week intervention
  Knee extensor fatigue will be assessed by a dynamometer.
Skeletal Muscle Cross Sectional Area | Change from baseline to after the 12 week intervention
  Skeletal muscle cross sectional area will be assessed via magnetic resonance imaging (MRI).
Skeletal Muscle Volume | Change from baseline to after the 12 week intervention
  Skeletal muscle volume will be assessed via magnetic resonance imaging (MRI).
Body Composition - Mass | Change from baseline to after the 12 week intervention
  Fat and fat free mass will be measured using by a dual x-ray absorptiometry (DEXA) scan.
Body Composition - Percentage | Change from baseline to after the 12 week intervention
  Fat and fat free percent will be measured using by a dual x-ray absorptiometry (DEXA) scan.
Skeletal Muscle Mitochondrial Respiration | Change from baseline to after the 12 week intervention
  Mitochondrial respiration will be assessed using high-resolution respirometry in permeabilized muscle fibers.
Skeletal Muscle Mitochondrial Hydrogen Peroxide Emissions | Change from baseline to after the 12 week intervention
  Mitochondrial hydrogen peroxide emissions will be assessed using high-resolution fluorometry in permeabilized muscle fibers.
Myofiber Size | Change from baseline to after the 12 week intervention
  Cross sectional area of muscle fibers will be evaluated with immunohistochemistry.

SECONDARY OUTCOMES:
Bone Density | Change from baseline to after the 12 week intervention
  Bone mineral density will be evaluated by a dual x-ray absorptiometry (DEXA) scan.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Konopka, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No